CLINICAL TRIAL: NCT01542476
Title: An Observational Study in Dutch Type 1 and Type 2 Diabetes Patients: The Impact of Initiation of/Switching to Levemir® on Emotional Well-being, Insulin Perceptions and Treatment Satisfaction - CONFIDENCE (Clinical ObservatioNs oF Levemir® In Dutch ExperieNCE)
Brief Title: The Impact of Initiating/Switching to Insulin Detemir on Emotional Well-being and Treatment Satisfaction
Acronym: CONFIDENCE
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN304-1924
Record Dates: First submitted 2012-02-24; First posted 2012-03-02 (Estimated); Last update posted 2016-03-03 (Estimated); Status verified 2016-03

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2 | interventions — Insulin Detemir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- IDet users
  Interventions: Drug: insulin detemir

INTERVENTIONS:
Drug: insulin detemir — Prescribed by the physician solely as a result of a normal clinical evaluation. The physician determines the starting dose and frequency, as well as later changes to either dose or frequency, if any

SUMMARY:
This study is conducted in Europe. The aim of this study is to assess the well-being of patients following treatment with insulin detemir (Levemir®) in subjects with type 1 or type 2 diabetes in whom either initiation of or a switch to insulin treatment with a long-acting basal insulin analogue is needed.

ELIGIBILITY:
Inclusion Criteria:

* Any subject with type 1 or type 2 diabetes not optimally controlled (HbA1c above 7.5%) in whom at the discretion of the participating physicians it was decide to either initiate or switch to a treatment with a long-acting insulin analogue
* Subjects with type 1 diabetes should have been treated with insulin for at least 12 months
* Potential pre-study treatment with insulin detemir (Levemir®) should have started no more than two months before baseline

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any subject with type 1 or type 2 diabetes not optimally controlled in whom at the discretion of the participating physicians it was decide to either initiate or switch to a treatment with a long-acting insulin analogue
Sampling Method: Non-Probability Sample
Enrollment: 299 (Actual)
Dates: Start 2006-08; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Change in Patient-Reported Outcomes (PRO) using World Health Organization 5 (WHO-5) item Well-being Index: Insulin Treatment Appraisal Scale (ITAS) | Baseline, month 6

SECONDARY OUTCOMES:
Change in Patient-Reported Outcomes (PRO) using Insulin Treatment (ITSQ) | Baseline, month 6
Change in HbA1c (glycosylated haemoglobin) | Baseline, month 6
Change in Fasting blood glucose (FBG) | Baseline, month 6
Change in body weight | Baseline, month 6
Hypoglycaemic episodes | Month 6
Adverse events | Month 6

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Alphen aan den Rijn, Netherlands

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com